CLINICAL TRIAL: NCT01689207
Title: A Phase I, Randomised, Double-blind, 3-Part Study in Healthy Young and Elderly Subjects to Assess the Safety and Tolerability, and Investigate the Pharmacokinetics of Aztreonam and Avibactam Given Alone and in Combination (ATM-AVI)
Brief Title: To Investigate the Safety and Tolerability of Aztreonam-Avibactam (ATM-AVI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4910C00001
Record Dates: First submitted 2012-09-12; First posted 2012-09-21 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Complicated Infection; Bacterial Infections
Keywords: Phase I, Safety, tolerability, healthy.
MeSH Terms: conditions — Bacterial Infections | interventions — avibactam; Aztreonam

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Drug: A (Experimental): Avibactam (AVI)
  Interventions: Drug: Avibactam (AVI)
- Drug: B (Experimental): Aztreonam (ATM)
  Interventions: Drug: Aztreonam (ATM)
- Drug: C (Experimental): combination of Aztreonam-Avibactam (ATM-AVI)
  Interventions: Drug: combination of Aztreonam - Avibactam (ATM-AVI)
- Drug: D (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avibactam (AVI) — PART A: AVI IV infusion
  Arms: Drug: A
Drug: Aztreonam (ATM) — PART A: ATM IV infusion
  Arms: Drug: B
Drug: combination of Aztreonam - Avibactam (ATM-AVI) — PART A: ATM-AVI IV infusion. PART B and C: ATM-AVI IV infusions.
  Arms: Drug: C
Drug: Placebo — PART A, PART B, PART C: matching placebo IV infusions
  Arms: Drug: D

SUMMARY:
This is a randomised, double-blind, 3-part study designed to investigate the safety and tolerability of ATM-AVI. The study aims to characterise the pharmacokinetics of ATM-AVI, when both drugs are administered alone (ATM or AVI) and in combination (ATM-AVI), following single administration, and following multiple administrations of ATM-AVI in healthy male and female (females of nonchildbearing potential) volunteers both young and elderly.

DETAILED DESCRIPTION:
A Phase I, Randomised, Double-blind, 3-Part Study in Healthy Young and Elderly Subjects to Assess the Safety and Tolerability, and Investigate the Pharmacokinetics of Aztreonam and Avibactam given Alone and in Combination (ATM-AVI)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy young male and female volunteers aged 18 to 45 years (inclusive) and healthy elderly volunteers aged 65 or older (Part C) with suitable veins for cannulation or repeated venipuncture
* Have a body mass index (BMI) between 19 and 30 kg/m2
* Be able to understand and willing to comply with study procedures, restrictions, and requirements, as judged by the PI

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Known history of severe allergy to betalactam and/or L-arginine
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to ATM or AVI
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks prior to the first administration of IP

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans van den Berg, MD, Principal Investigator — Hammersmith Medicines Research Cumberland Avenue Park Royal London NW10 7EW, England Telephone: +44 020 8961 4130 Fax: +44 020 8961 8665
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Das S, Riccobene T, Carrothers TJ, Wright JG, MacPherson M, Cristinacce A, McFadyen L, Xie R, Luckey A, Raber S. Dose selection for aztreonam-avibactam, including adjustments for renal impairment, for Phase IIa and Phase III evaluation. Eur J Clin Pharmacol. 2024 Apr;80(4):529-543. doi: 10.1007/s00228-023-03609-x. Epub 2024 Jan 22. PMID 38252170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 27 September 2012 and last subject last visit was 30 December 2014. Subjects were healthy male and female volunteers both young and elderly. Healthy volunteers were given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study and could discontinue at any time.
Pre-assignment Details: A Screening visit was conducted within 28 days before admission to the study centre. 222 volunteers were screend, 92 volunteers were entered into the study. Healthy volunteers were admitted to the study centre on Day -1 of either Part A, Part B or Part C.
Groups:
- Part A: Placebo; Part B: Placebo; Part C: Placebo: Placebo
- Part A: Drug: Aztreonam (ATM) 2000mg, Avibactam (AVI) 600mg, ATM 2000mg +AVI 600mg (crossover)
- Part B: Cohort 1 Drug: ATM (2000mg) + AVI (375mg)
- Part B: Cohort 2 Drug: ATM (2000mg) + AVI (600mg)
- Part B: Cohort 3 Drug: ATM (1500mg) + AVI (600mg)
- Part B: Cohort 4 Drug: ATM (1500mg) + AVI (450mg)
- Part B: Cohort 5 Drug: ATM (1500mg) + AVI (410mg)
- Part C: Cohort 1 Drug: Aged 18-45: ATM (500mg followed by 1500mg) + AVI (136.7mg followed by 410mg)
- Part C: Cohort 2 Drug: Aged >65: ATM (500mg followed by 1500mg) + AVI (136.7mg + 410mg)
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug
Started | 4 (Subjects randomised) | 8 (Subjects randomised) | 16 (Subjects randomised) | 8 (Subjects randomised) | 4 (Subjects randomised) | 8 (Subjects randomised) | 10 (Subjects randomised) | 10 (Subjects randomised) | 6 (Subjects randomised) | 10 (Subjects randomised) | 8 (Subjects randomised)
Completed | 4 (Subjects completed study) | 7 (Subjects completed study) | 16 (Subjects completed study) | 8 (Subjects completed study) | 2 (Subjects completed study) | 7 (Subjects completed study) | 10 (Subjects completed study) | 10 (Subjects completed study) | 5 (Subjects completed study) | 10 (Subjects completed study) | 8 (Subjects completed study)
Not Completed | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomised subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug | Total
Number analyzed (Participants) | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 6 | 10 | 8 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (6.9) | 31.3 (7.1) | 27.4 (5.0) | 30.3 (4.9) | 27.8 (1.9) | 29.4 (9.9) | 29.7 (7.3) | 30.6 (6.3) | 51.3 (19.4) | 32.9 (8.4) | 68.5 (2.9) | 34.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Male | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 5 | 10 | 6 | 89

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile - Number of Subjects With at Least 1 AE
Description: from screening visit (Day -28) to 3 to 7 days post treatment period 3 (up to Day 22) in Part A, 3 to 7 days after receiving the final dose on Day 11 (days 14 to 18) in Part B, and 3 to 7 days after receiving the final dose on Day 10 (days 13 to 17) in Part C.
Time Frame: Informed consent (up to 28 days before first dose) to follow up period (max of 22 days after first dose for Part A, a max of 28 days after first dose in Part B, max 17 days in Part C)
Population: Safety population
Measure: Number; unit: Participants
Groups:
- Part A: Aztreonam (ATM) 2000mg: Crossover period ATm 2000mg
- Part A: Avibactam (AVI) 600mg: Crossover period AVI 600mg
- Part A: ATM 2000mg + AVI 600mg: Crossover period ATM 2000mg + AVI 600mg
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug | Part A: Aztreonam (ATM) 2000mg | Part A: Avibactam (AVI) 600mg | Part A: ATM 2000mg + AVI 600mg
Number analyzed (Participants) | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 6 | 10 | 8 | 7 | 8 | 7
Participants
  Number of subjects with at least 1 AE | 1 | 2 | 3 | 4 | 2 | 6 | 8 | 3 | 3 | 5 | 7 | 0 | 2 | 0
  Subjects with at least 1 AE with outcome of death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least 1 AE leading to discontinuation | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: PK- Plasma Pharmacokinetic Parameter AUC (ug*h/mL) for Aztreonam (ATM) and Avibactam (AVI) Alone and in Combination (ATM-AVI) in Parts A, B and C
Description: Area under the plasma concentration-time curve from zero extrapolated to infinity (AUC µg*h/mL) or AUC(0-last) in Part A on Day 1 after single infusion, area under the plasma concentration-time curve at steady state after multiple infusion (AUCss µg*h/mL).
Time Frame: 0 to 24 hours post-dose on Day 1 in Part A. 0 to 24 hours post-dose on Days 1, 2, 4 and 11 in Part B (varied intervals per cohort). 0 to 6 hours post-dose on Days 1, 4, 7 and 10 in Part C. Steady state measure on Day 11 in Part B or Day 10 in Part C
Population: Pharmacokinetic analysis set. Please note, PK parameters have not been calculated where data is available in <3 subjects as this is considered to lack robustness.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug
Number analyzed (Participants) | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 6 | 10 | 8
ug*h/mL
  AUC (ug*h/mL) - Aztreonam (ATM) alone | NA (NA) — Not evaluated | 372 (15.2) | NA (NA) — Not evaluated | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone | NA (NA) — Not evaluated | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone
  AUC (ug*h/mL) - Avibactam (AVI)alone | NA (NA) — Not evaluated | 52.6 (22.5) | NA (NA) — Not evaluated | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone | NA (NA) — Not evaluated | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone
  AUC (ug*h/mL) - ATM in combination (Day 1) | NA (NA) — Not evaluated | 375 (12.8) | NA (NA) — Not evaluated | 345 (16.3) | 326 (5.5) | 283 (17.7) | 270 (9.8) | 250 (13.3) | NA (NA) — Not evaluated | 276 (13.5) | 308 (12.0)
  AUCss (ug*h/mL) - ATM in combination | NA (NA) — Not evaluated | NA (NA) — No multiple dosing | NA (NA) — Not evaluated | 275 (14.0) | NA (NA) — Not determined as only 2 subjects | 231 (15.9) | 223 (7.9) | 203 (11.1) | NA (NA) — Not evaluated | 211 (15.7) | 259 (12.1)
  AUC (ug*h/mL) - AVI in combination (Day 1) | NA (NA) — Not evaluated | 58.3 (17.7) | NA (NA) — Not evaluated | 31.8 (12.5) | 47.8 (12.5) | 53.1 (12.9) | 35.7 (11.8) | 31.4 (14.7) | NA (NA) — Not evaluated | 41.9 (17.1) | 52.3 (11.0)
  AUCss (ug*h/mL) - AVI in combination | NA (NA) — Not evaluated | NA (NA) — No multiple dosing in Part A | NA (NA) — Not evaluated | 26.1 (13.0) | NA (NA) — Not determined as only 2 subjects | 43.3 (11.7) | 29.0 (10.2) | 26.7 (12.6) | NA (NA) — Not evaluated | 29.3 (19.6) | 38.8 (14.0)

3. Secondary Outcome: PK- Plasma Pharmacokinetic Parameter t1/2(h) for Aztreonam (ATM) and Avibactam (AVI) Alone and in Combination (ATM-AVI) in Parts A, B and C
Description: Terminal half-life (t1/2), on Day 1 after single infusion and at steady state after multiple infusion.
Time Frame: as for outcome 2
Population: Pharmacokinetic analysis set. Please note, PK parameters have not been calculated where data is available in <3 subjects as this is considered to lack robustness. Placebo arms are not evaluated. Values shown where analysed (eg. not applicable for ATM alone in combination cohorts)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug
Number analyzed (Participants) | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 6 | 10 | 8
h
  t1/2 (h) - Aztreonam (ATM) alone | NA (NA) — Not evaluated | 1.98 (18.9) | NA (NA) — Not evaluated | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — Not evaluated | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone
  t1/2 (h) - Avibactam (AVI)alone | NA (NA) — Not evaluated | 2.22 (26.3) | NA (NA) — Not evaluated | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — Not evaluated | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone
  t1/2 (h) - ATM in combination | NA (NA) — Not evaluated | 2.09 (14.0) | NA (NA) — Not evaluated | 2.24 (16.6) | 1.98 (3.3) | 1.90 (16.2) | 2.14 (21.2) | 2.28 (25.9) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated
  t1/2 (h) - AVI in combination | NA (NA) — Not evaluated | 2.35 (25.4) | NA (NA) — Not evaluated | 2.17 (30.9) | 2.82 (41.1) | 2.61 (10.1) | 2.26 (30.1) | 1.85 (27.4) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated

4. Secondary Outcome: PK- Plasma Pharmacokinetic Parameter Tmax for Aztreonam (ATM) and Avibactam (AVI) Alone and in Combination (ATM-AVI) on Day 1 in Parts A, B and C
Description: Time to Cmax (tmax)
Time Frame: Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: (h)
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug
Number analyzed (Participants) | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 6 | 10 | 8
(h)
  tmax (h) - ATM alone | NA [NA to NA] — Not evaluated | 0.98 [0.98 to 0.98] | NA [NA to NA] — Not evaluated | NA [NA to NA] — ATM not dosed alone | NA [NA to NA] — ATM not dosed alone | NA [NA to NA] — ATM not dosed alone | NA [NA to NA] — ATM not dosed alone | NA [NA to NA] — ATM not dosed alone | NA [NA to NA] — Not evaluated | NA [NA to NA] — ATM not dosed alone | NA [NA to NA] — ATM not dosed alone
  tmax (h) - AVI alone | NA [NA to NA] — Not evaluated | 0.98 [0.98 to 1.12] | NA [NA to NA] — Not evaluated | NA [NA to NA] — AVI not dosed alone | NA [NA to NA] — AVI not dosed alone | NA [NA to NA] — AVI not dosed alone | NA [NA to NA] — AVI not dosed alone | NA [NA to NA] — AVI not dosed alone | NA [NA to NA] — Not evaluated | NA [NA to NA] — AVI not dosed alone | NA [NA to NA] — AVI not dosed alone
  tmax (h) - ATM in combination (Day 1) | NA [NA to NA] — Not evaluated | 0.98 [0.98 to 0.98] | NA [NA to NA] — Not evaluated | 0.98 [0.98 to 1.25] | 0.98 [0.98 to 1.00] | 1.98 [1.50 to 1.98] | 2.98 [2.00 to 3.00] | 2.98 [2.50 to 3.03] | NA [NA to NA] — Not evaluated | 2.98 [2.98 to 3.00] | 2.98 [2.68 to 3.03]
  tmax (h) - AVI in combination (Day 1) | NA [NA to NA] — Not evaluated | 0.98 [0.98 to 0.98] | NA [NA to NA] — Not evaluated | 0.98 [0.98 to 0.98] | 0.98 [0.98 to 1.00] | 1.98 [1.50 to 1.98] | 2.98 [2.00 to 3.00] | 2.50 [2.50 to 3.05] | NA [NA to NA] — Not evaluated | 2.98 [2.00 to 3.00] | 2.98 [2.50 to 3.03]

5. Secondary Outcome: PK- Plasma Pharmacokinetic Parameter Cmax for Aztreonam (ATM) and Avibactam (AVI) Alone and in Combination (ATM-AVI) in Parts A, B and C
Description: Maximum plasma concentration (Cmax µg/mL) on Day 1 after single infusion , maximum plasma concentration at steady state (Css,max µg/mL) after multiple infusion.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug
Number analyzed (Participants) | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 6 | 10 | 8
ug/mL
  Cmax (ug/mL) - ATM alone | NA (NA) — Not evaluated | 143 (14.0) | NA (NA) — Not evaluated | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone | NA (NA) — Not evaluated | NA (NA) — ATM not administered alone | NA (NA) — ATM not administered alone
  Cmax (ug/mL) - AVI alone | NA (NA) — Not evaluated | 26.8 (14.2) | NA (NA) — Not evaluated | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone | NA (NA) — Not evaluated | NA (NA) — AVI not administered alone | NA (NA) — AVI not administered alone
  Cmax (ug/mL) - ATM in combination (Day1) | NA (NA) — Not evaluated | 137 (11.3) | NA (NA) — Not evaluated | 123 (16.7) | 123 (6.2) | 82.4 (16.0) | 63.2 (9.4) | 59.2 (13.1) | NA (NA) — Not evaluated | 75.6 (13.8) | 81.6 (11.8)
  Css, max (ug/mL) - ATM in combination | NA (NA) — Not evaluated | NA (NA) — No multiple dosing in Part A | NA (NA) — Not evaluated | 124 (9.0) | NA (NA) — Not determined as only 2 subjects | 80.9 (12.9) | 62.6 (9.1) | 55.7 (9.0) | NA (NA) — Not evaluated | 57.2 (14.9) | 66.2 (13.3)
  Cmax (ug/mL) - AVI in combination (Day1) | NA (NA) — Not evaluated | 137 (11.3) | NA (NA) — Not evaluated | 16.0 (10.1) | 25.1 (5.8) | 19.3 (16.4) | 9.99 (11.2) | 8.68 (14.0) | NA (NA) — Not evaluated | 12.1 (18.4) | 15.2 (13.6)
  Css, max (ug/mL) - AVI in combination | NA (NA) — Not evaluated | NA (NA) — No multiple dosing in Part A | NA (NA) — Not evaluated | 14.5 (15.9) | NA (NA) — Not determined as only 2 subjects | 17.6 (12.2) | 8.69 (9.9) | 8.36 (16.5) | NA (NA) — Not evaluated | 8.88 (19.9) | 11.6 (15.1)

6. Secondary Outcome: PK- Plasma Pharmacokinetic Parameters CL and CLr for Aztreonam (ATM) and Avibactam (AVI) Alone and in Combination (ATM-AVI) in Parts A, B and C
Description: Systemic clearence (CL) and renal clearance (CLr) on Day 1 after single infusion and at steady state after multiple infusion.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug
Number analyzed (Participants) | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 6 | 10 | 8
L/h
  CL (L/h) - ATM alone | NA (NA) — Not evaluated | 5.37 (15.2) | NA (NA) — Not evaluated | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — Not evaluated | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone
  CL(L/h) - AVI alone | NA (NA) — Not evaluated | 11.4 (22.4) | NA (NA) — Not evaluated | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — Not evaluated | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone
  CLr (L/h) - ATM alone | NA (NA) — Not evaluated | 3.93 (19.0) | NA (NA) — Not evaluated | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — Not evaluated | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone
  CLr (L/h) - AVI alone | NA (NA) — Not evaluated | 9.77 (21.6) | NA (NA) — Not evaluated | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — Not evaluated | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone
  CL(L/h) - ATM in combination (Day 1) | NA (NA) — Not evaluated | 5.33 (12.9) | NA (NA) — Not evaluated | 5.79 (16.3) | 6.15 (5.5) | 5.29 (17.8) | 5.56 (9.9) | 5.99 (13.4) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated
  CLr (L/h) - ATM in comination (Day 1) | NA (NA) — Not evaluated | 3.78 (17.6) | NA (NA) — Not evaluated | 4.04 (14.4) | 4.10 (7.4) | 4.18 (14.0) | 4.09 (21.5) | 4.43 (11.8) | NA (NA) — Not evaluated | 4.22 (17.2) | 3.41 (16.9)
  CL(L/h) - AVI in combination (Day 1) | NA (NA) — Not evaluated | 10.3 (17.7) | NA (NA) — Not evaluated | 11.8 (12.4) | 12.5 (12.7) | 11.3 (12.8) | 12.6 (11.9) | 13.1 (14.8) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated
  CLr (L/h) - AVI in comination (Day 1) | NA (NA) — Not evaluated | 8.71 (17.1) | NA (NA) — Not evaluated | 10.6 (19.3) | 10.9 (12.5) | 11.1 (11.7) | 11.9 (24.6) | 12.5 (15.6) | NA (NA) — Not evaluated | 10.8 (16.3) | 7.78 (27.9)
  CL(L/h) - ATM in combination (Steady state) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated | 7.27 (14.0) | NA (NA) — Not calculated as <3 patients | 6.49 (15.9) | 6.72 (7.9) | 7.39 (11.1) | NA (NA) — Not evaluated | 7.10 (15.8) | 5.79 (12.2)
  CLr (L/h) - ATM in comination (Steady state) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated | 4.66 (18.9) | NA (NA) — Not calculated as <3 patients | 4.93 (15.2) | 5.07 (27.8) | 5.25 (13.5) | NA (NA) — Not evaluated | 4.97 (19.0) | 3.99 (21.0)
  CL(L/h) - AVI in combination (Steady state) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated | 14.3 (13.1) | NA (NA) — Not calculated as <3 patients | 13.8 (11.7) | 15.5 (10.4) | 15.4 (12.7) | NA (NA) — Not evaluated | 14.0 (19.7) | 10.6 (14.0)
  CLr (L/h) - AVI in comination (Steady state) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated | 12.4 (24.8) | NA (NA) — Not calculated as <3 patients | 13.9 (11.5) | 14.7 (24.6) | 14.5 (14.6) | NA (NA) — Not evaluated | 13.0 (22.0) | 9.49 (18.7)

7. Secondary Outcome: PK- Plasma Pharmacokinetic Parameter Vss for Aztreonam (ATM) and Avibactam (AVI) Alone and in Combination (ATM-AVI) in Parts A, B and C
Description: Volume of distribution at steady state (Vss).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug
Number analyzed (Participants) | 4 | 8 | 16 | 8 | 4 | 8 | 10 | 10 | 6 | 10 | 8
L
  Vss (L) - ATM alone | NA (NA) — Not evaluated | 13.4 (16.3) | NA (NA) — Not evaluated | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone | NA (NA) — Not evaluated | NA (NA) — ATM not dosed alone | NA (NA) — ATM not dosed alone
  Vss (L) - AVI alone | NA (NA) — Not evaluated | 20.1 (10.0) | NA (NA) — Not evaluated | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone | NA (NA) — Not evaluated | NA (NA) — AVI not dosed alone | NA (NA) — AVI not dosed alone
  Vss (L) - ATM in comination | NA (NA) — Not evaluated | 13.8 (10.4) | NA (NA) — Not evaluated | 15.4 (13.3) | 15.1 (5.2) | 12.5 (14.9) | 13.7 (11.9) | 15.6 (18.9) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated
  Vss (L) - AVI in comination | NA (NA) — Not evaluated | 19.0 (15.3) | NA (NA) — Not evaluated | 22.8 (15.6) | 22.2 (10.6) | 20.0 (18.9) | 23.5 (15.5) | 25.2 (26.0) | NA (NA) — Not evaluated | NA (NA) — Not evaluated | NA (NA) — Not evaluated

ADVERSE EVENTS:
Time Frame: from screening visit (Day -28) to follow up visit (FUP).
Description: FUP=3 to 7 days post treatment period 3 (up to Day 22) in Part A, 3 to 7 days after receiving the final dose on Day 11 (days 14 to 18) in Part B, and 3 to 7 days after receiving the final dose on Day 10 (days 13 to 17) in Part C.
Arm/Group | Part A: Placebo | Part A: Drug | Part B: Placebo | Part B: Cohort 1 Drug | Part B: Cohort 2 Drug | Part B: Cohort 3 Drug | Part B: Cohort 4 Drug | Part B: Cohort 5 Drug | Part C: Placebo | Part C: Cohort 1 Drug | Part C: Cohort 2 Drug | Part A: Aztreonam (ATM) 2000mg | Part A: Avibactam (AVI) 600mg | Part A: ATM 2000mg + AVI 600mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 0/16 | 0/8 | 0/4 | 0/8 | 0/10 | 0/10 | 1/6 | 0/10 | 0/8 | 0/7 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/4 | 2/8 | 3/16 | 4/8 | 2/4 | 6/8 | 8/10 | 3/10 | 3/6 | 5/10 | 7/8 | 0/7 | 2/8 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=4) | Part A: Drug (N=8) | Part B: Placebo (N=16) | Part B: Cohort 1 Drug (N=8) | Part B: Cohort 2 Drug (N=4) | Part B: Cohort 3 Drug (N=8) | Part B: Cohort 4 Drug (N=10) | Part B: Cohort 5 Drug (N=10) | Part C: Placebo (N=6) | Part C: Cohort 1 Drug (N=10) | Part C: Cohort 2 Drug (N=8) | Part A: Aztreonam (ATM) 2000mg (N=7) | Part A: Avibactam (AVI) 600mg (N=8) | Part A: ATM 2000mg + AVI 600mg (N=7)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=4) | Part A: Drug (N=8) | Part B: Placebo (N=16) | Part B: Cohort 1 Drug (N=8) | Part B: Cohort 2 Drug (N=4) | Part B: Cohort 3 Drug (N=8) | Part B: Cohort 4 Drug (N=10) | Part B: Cohort 5 Drug (N=10) | Part C: Placebo (N=6) | Part C: Cohort 1 Drug (N=10) | Part C: Cohort 2 Drug (N=8) | Part A: Aztreonam (ATM) 2000mg (N=7) | Part A: Avibactam (AVI) 600mg (N=8) | Part A: ATM 2000mg + AVI 600mg (N=7)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
No formal statistical hypothesis testing was performed. The analyses of safety, tolerability, and pharmacokinetic data were summarised descriptively including tables, listings, and graphs, as appropriate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality clauses are in place through a Master Services agreement, which limits the discloser of confidential information to what's expressed in 33.2 and 33.3: disclosure to third party only after written consent, or disclosure of confidential information only to the extent necessary to comply with reporting obligations from AZ, CRO or applicable laws.